CLINICAL TRIAL: NCT00620971
Title: Sequential Cisplatin/Vinorelbine/Bevacizumab Followed by Docetaxel/Gemcitabine/Bevacizumab Versus Cisplatin/Docetaxel/Bevacizumab in Patients With Locally Advanced or Metastatic Non Small Cell Lung Cancer
Brief Title: Cisplatin/Vinorelbine/Bevacizumab Followed by Docetaxel/Gemcitabine/Bevacizumab Versus the Cisplatin/Docetaxel/Bevacizumab Combination in Locally Advanced or Metastatic NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/07.19
Record Dates: First submitted 2008-01-31; First posted 2008-02-22 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Cisplatin; VInorelbine; Docetaxel; Gemcitabine; Bevacizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vinorelbine; Cisplatin; Bevacizumab; Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): NC/Avastin->DG/Avastin
  Interventions: Drug: Vinorelbine; Drug: Cisplatin; Drug: Bevacizumab; Drug: Docetaxel; Drug: Gemcitabine
- 2 (Experimental): DG/Avastin
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Vinorelbine — Vinorelbine (oral) 60 mg/m2, on days 1 and 8 every 3 weeks for 3 cycles
  Other Names: Navelbine
  Arms: 1
Drug: Cisplatin — Cisplatin (IV) 80 mg/m2 on day 1 every 3 weeks for 3 cycles
  Other Names: CDDP
  Arms: 1
Drug: Bevacizumab — Bevacizumab (IV) 15 mgr/Kgr on day 1 every 3 weeks for 3 cycles
  Other Names: Avastin
  Arms: 1
Drug: Docetaxel — Docetaxel (IV) 75 mg/m2 on day 1 every 3 weeks for 6 cycles
  Other Names: Taxotere
  Arms: 1
Drug: Gemcitabine — Gemcitabine(IV) 1,100 mg/m2 on day 1 and d8 every 3 weeks for 6 cycles
  Other Names: Gemzar
  Arms: 1
Drug: Bevacizumab — Bevacizumab (IV) 15 mgr/Kgr on day 1 every 3 weeks for 6 cycles
  Other Names: Avastin
  Arms: 1
Drug: Docetaxel — Docetaxel (IV) 75 mg/m2 on day 1 every 3 weeks for 6 cycles
  Other Names: Taxotere
  Arms: 2
Drug: Cisplatin — Cisplatin (IV) 80 mg/m2 on day 1 every 3 weeks for 6 cycles
  Other Names: CDDP
  Arms: 2
Drug: Bevacizumab — Bevacizumab (IV) 15 mgr/Kgr on day 1 every 3 weeks for 6 cycles
  Other Names: Avastin
  Arms: 2

SUMMARY:
This trial will evaluate whether the sequential administration of Cisplatin/Vinorelbine/Bevacizumab followed by Docetaxel/Gemcitabine/Bevacizumab versus the Cisplatin/Docetaxel/Bevacizumab combination as first line treatment offers a survival advantage in patients with locally advanced or metastatic NSCLC.

DETAILED DESCRIPTION:
An unanswered question in first line treatment of non small cell lung cancer (NSCLC) is whether the administration of more than 2 active drugs provides greater efficacy than a two-drug combination. Docetaxel/gemcitabine combination is a well tolerated regimen, which has comparable efficacy to docetaxel/cisplatin or vinorelbine/cisplatin. In a recent phase II study in first line treatment of advanced or metastatic NSCLC, the sequential administration of vinorelbine/cisplatin followed by docetaxel/gemcitabine produced a response rate of 45.8% and a 1-year survival rate of 51%. The addition of bevacizumab to a platinum-based regimen provided a survival benefit in patients with advanced or metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, unresectable locally advanced (stage IIIB with pleural effusion) or metastatic (stage IV) non-squamous NSCLC
* Performance status (WHO) 0-1
* Adequate bone marrow (ANC ≥ 1,500/mm3, PLT ≥ 100,000/mm3, Hgb ≥ 11 g/dL), liver (Bilirubin ≤ 1.5 UNL, SGOT/SGPT ≤ 2.5 UNL, ALP ≤ 5 UNL), and renal function (Creatinine ≤ UNL - if borderline, creatinine clearance should be ≥ 60 mL/min)
* No previous chemotherapy or immunotherapy for advanced/metastatic NSCLC is allowed

  --Previous radiotherapy is allowed provided that the measurable lesions are outside the radiation fields
* Measurable disease, defined as at least 1 bidimensionally measurable lesion ≥ 20 X 10 mm
* Patient able to take oral medication
* Absence of active CNS disease
* Paraffin embedded sample of primary or metastatic tumor diagnostic specimen must be available
* Patients must be able to understand the nature of this study and give written informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Women of child-bearing age unable or unwilling to take effective contraceptive measures
* Active CNS disease, brain metastases, or leptomeningeal involvement
* Symptomatic neuropathy > grade1 according to the NCI CTCAE (version 3.0)
* Cardiovascular disease (class II-IV NYHA congestive heart failure, myocardial infarction within the previous 4 months, LVEF < normal, uncontrolled hypertension, ventricular arrhythmia), anticoagulation treatment or thrombotic event within the previous 6 months
* Active infection, requiring IV antibiotic treatment, within the previous 2 weeks
* Long-term oxygen therapy
* Second primary malignancy, except for non-melanoma skin cancer and in situ cervical cancer
* Radiotherapy within the previous 4 weeks
* Previous radiotherapy to the only measurable lesion
* Concurrent treatment with other anti-cancer drug
* Uncontrolled hypercalcemia
* Known allergy to drugs with similar chemical structure to study drugs. Concurrent corticosteroids, except for chronic therapy with methylprednisolone ≤ 20 mgr daily (or equivalent) for more than one month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)

SECONDARY OUTCOMES:
Time to Tumor Progression | 1-year
Overall Survival | 1 year
Quality of life assessment | Assessment every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (9):
- Greece (9):
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - "Metaxa's" Anticancer Hospital of Piraeus,1st Dep of Medical Oncology, Athens
  - 401 Military Hospital, Medical Oncology Unit, Athens
  - Air Forces Military Hospital, Dep of Medical Oncology, Athens
  - IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - Sismanogleio General Hospital, 1st, 2nd Dep of Pulmonary Diseases, Athens
  - Sotiria" General Hospital, 1st, 3rd, 8th Dep of Pulmonary Diseases, Athens
  - "Theagenion" Anticancer Hospital of Thessaloniki, Thessaloniki

REFERENCES:
- [Derived] Kotsakis A, Kentepozidis N, Emmanouilidis Ch, Polyzos A, Agelidou A, Vaslamatzis M, Chandrinos V, Agelaki S, Vamvakas L, Kalbakis K, Katsaounis P, Stoltidis D, Nintos G, Hatzidaki D, Vetsika EK, Mavroudis D, Georgoulias V. Sequential administration of vinorelbine plus cisplatin and bevacizumab followed by docetaxel plus gemcitabine and bevacizumab compared to docetaxel plus cisplatin and bevacizumab regimen as first-line therapy for advanced or metastatic non-squamous non-small cell lung cancer: A multicenter randomized phase II trial of the Hellenic Oncology Research Group (HORG). Lung Cancer. 2015 Apr;88(1):57-62. doi: 10.1016/j.lungcan.2015.01.012. Epub 2015 Jan 23. PMID 25662596